CLINICAL TRIAL: NCT00934752
Title: An Exploratory Study Investigating the Use of the Lutonix Paclitaxel-Coated Balloon in Conjunction With Bare Metal Stenting in Patients With De Novo Coronary Lesions.
Brief Title: De Novo Pilot Study, Lutonix Catheter in Conjunction With Bare Metal Stenting for Treatment of Coronary De Novo Lesions
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL0013-01
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Coronary Artery Stenosis
Keywords: de novo stenotic lesions
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lutonix Catheter (Experimental)
  Interventions: Device: Lutonix Paclitaxel-Coated Balloon

INTERVENTIONS:
Device: Lutonix Paclitaxel-Coated Balloon — Percutaneous transluminal coronary angioplasty (PCTA)
  Other Names: Drug Coated Balloon

SUMMARY:
The study will enroll patients with angiographically significant coronary de novo lesions. Subjects will be randomized 1:1 and treated with a Lutonix catheter either before or after bare-metal stenting (BMS). The purpose is to assess the feasibility, safety and efficacy of the Lutonix Catheter for treatment of de novo coronary artery stenosis using two distinct treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant/non-breast feeding Female ≥ 18 years of age. Women of childbearing potential must have a negative pregnancy test (within 7 days of the procedure);
* Documented stable angina pectoris Canadian Cardiovascular Society Classification (CCSC) 1-4, unstable angina pectoris with documented ischemia (Braunwald I-II) or documented silent ischemia;
* Left ventricular ejection fraction (LVEF) ≥ 25%;
* Patient is an acceptable candidate for PTCA, stenting, and emergent coronary artery bypass grafting (CABG);
* Patient is willing to provide informed consent and comply with follow-up visits and testing schedule;
* Target lesion is a de novo lesion in a native coronary artery vessel;
* Initial stenosis is ≥ 50% and < 100% by visual estimate or quantitative coronary angiography (QCA);
* Reference Vessel Diameter (RVD) is ≥ 2.5 and ≤ 3.25 prior to predilation;
* Target lesion is ≤18mm in length and can be treated in its entirety by no more than 1 single Lutonix Catheter balloon and 1 single BMS;
* Guidewire is able to cross lesion and be placed in distal vessel prior to enrollment;
* Enrollment permitted after successful treatment of 1 non-study lesion in a single other non-study vessel (not in the same vascular territory as the study lesion). Successful treatment is defined as ≤ 30% residual stenosis with Thrombolysis in Myocardial Infarction (TIMI) Grade III flow and not evidence of dissection.

Exclusion Criteria:

* History of stroke within past 6 months;
* History of myocardial infarction (MI) or thrombolysis within 72 hours of randomization;
* Prior vascular brachytherapy;
* Uncontrollable allergies to procedure medications, materials or contrast;
* Angiographic evidence of thrombus or dissection within the target vessel;
* Intervention of another coronary lesion ≤ 60 days before index procedure day or planned following index procedure;
* Target lesion is planned to be treated with something other than PTCA and stent (i.e., cutting-balloon, atherectomy, vascular brachytherapy (VBT), etc.);
* Target lesion is in the Left Main and has excessive calcification or tortuosity or involves bifurcation disease of vessel ≥ 2.5mm;
* Known sensitivity or has received paclitaxel or other antimitogenic agent within 12 months prior to target vessel treatment;
* Patient has any previous intervention (PTCA, stent, etc.) of the target coronary vessel;
* Any medical condition, in the investigators opinion, that should preclude the patient from the study or patient has a life expectancy less than 24 months;
* Known creatine kinase-MB (CKMB) > 2x upper limit of normal (ULN) or positive Troponin;
* Creatinine > 2.0 mg/dl;
* Leukocyte < 3500/mL;
* Platelet < 100,000 mL or > 750,000 mL;
* Currently taking or must resume warfarin;
* Patient is contraindicated for antiplatelet therapy or it will need to be withdrawn for a planned procedure;
* The subject is currently participating in another investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Mean percent stent volume obstruction as measured by optical coherence tomography (OCT) | 6 months

SECONDARY OUTCOMES:
Stent Malposition | 6 Months
Minimal Lumen Area | 6 Months
Stent Symmetry | 6 Months
Stent Expansion | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Prof. P.W.J C. Serruys, MD, PhD, Principal Investigator — Erasmus Universtiy Medical Center; Netherlands
Locations (3):
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - Catherina Zeikenhuis, Eindhoven
  - Thorax Center, Rotterdam

REFERENCES:
- [Background] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Background] Colombo A, Drzewiecki J, Banning A, Grube E, Hauptmann K, Silber S, Dudek D, Fort S, Schiele F, Zmudka K, Guagliumi G, Russell ME; TAXUS II Study Group. Randomized study to assess the effectiveness of slow- and moderate-release polymer-based paclitaxel-eluting stents for coronary artery lesions. Circulation. 2003 Aug 19;108(7):788-94. doi: 10.1161/01.CIR.0000086926.62288.A6. Epub 2003 Aug 4. PMID 12900339
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Eisenstein EL, Anstrom KJ, Kong DF, Shaw LK, Tuttle RH, Mark DB, Kramer JM, Harrington RA, Matchar DB, Kandzari DE, Peterson ED, Schulman KA, Califf RM. Clopidogrel use and long-term clinical outcomes after drug-eluting stent implantation. JAMA. 2007 Jan 10;297(2):159-68. doi: 10.1001/jama.297.2.joc60179. Epub 2006 Dec 5. PMID 17148711
- [Background] Acute platelet inhibition with abciximab does not reduce in-stent restenosis (ERASER study). The ERASER Investigators. Circulation. 1999 Aug 24;100(8):799-806. doi: 10.1161/01.cir.100.8.799. PMID 10458714
- [Background] Erbel R, Haude M, Hopp HW, Franzen D, Rupprecht HJ, Heublein B, Fischer K, de Jaegere P, Serruys P, Rutsch W, Probst P. Coronary-artery stenting compared with balloon angioplasty for restenosis after initial balloon angioplasty. Restenosis Stent Study Group. N Engl J Med. 1998 Dec 3;339(23):1672-8. doi: 10.1056/NEJM199812033392304. PMID 9834304
- [Background] Fischman DL, Leon MB, Baim DS, Schatz RA, Savage MP, Penn I, Detre K, Veltri L, Ricci D, Nobuyoshi M, et al. A randomized comparison of coronary-stent placement and balloon angioplasty in the treatment of coronary artery disease. Stent Restenosis Study Investigators. N Engl J Med. 1994 Aug 25;331(8):496-501. doi: 10.1056/NEJM199408253310802. PMID 8041414
- [Background] Gonzalo N, Garcia-Garcia HM, Serruys PW, Commissaris KH, Bezerra H, Gobbens P, Costa M, Regar E. Reproducibility of quantitative optical coherence tomography for stent analysis. EuroIntervention. 2009 Jun;5(2):224-32. doi: 10.4244/eijv5i2a35. PMID 19527980
- [Background] Holmes DR Jr, Teirstein P, Satler L, Sketch M, O'Malley J, Popma JJ, Kuntz RE, Fitzgerald PJ, Wang H, Caramanica E, Cohen SA; SISR Investigators. Sirolimus-eluting stents vs vascular brachytherapy for in-stent restenosis within bare-metal stents: the SISR randomized trial. JAMA. 2006 Mar 15;295(11):1264-73. doi: 10.1001/jama.295.11.1264. Epub 2006 Mar 12. PMID 16531619
- [Background] Joner M, Finn AV, Farb A, Mont EK, Kolodgie FD, Ladich E, Kutys R, Skorija K, Gold HK, Virmani R. Pathology of drug-eluting stents in humans: delayed healing and late thrombotic risk. J Am Coll Cardiol. 2006 Jul 4;48(1):193-202. doi: 10.1016/j.jacc.2006.03.042. Epub 2006 May 5. PMID 16814667
- [Background] King SB 3rd, Smith SC Jr, Hirshfeld JW Jr, Jacobs AK, Morrison DA, Williams DO, Feldman TE, Kern MJ, O'Neill WW, Schaff HV, Whitlow PL; ACC/AHA/SCAI; Adams CD, Anderson JL, Buller CE, Creager MA, Ettinger SM, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Page RL, Riegel B, Tarkington LG, Yancy CW. 2007 focused update of the ACC/AHA/SCAI 2005 guideline update for percutaneous coronary intervention: a report of the American College of Cardiology/American Heart Association Task Force on Practice guidelines. J Am Coll Cardiol. 2008 Jan 15;51(2):172-209. doi: 10.1016/j.jacc.2007.10.002. No abstract available. PMID 18191745
- [Background] Lee MS, Pessegueiro A, Zimmer R, Jurewitz D, Tobis J. Clinical presentation of patients with in-stent restenosis in the drug-eluting stent era. J Invasive Cardiol. 2008 Aug;20(8):401-3. PMID 18688064
- [Background] Mauri L, Hsieh WH, Massaro JM, Ho KK, D'Agostino R, Cutlip DE. Stent thrombosis in randomized clinical trials of drug-eluting stents. N Engl J Med. 2007 Mar 8;356(10):1020-9. doi: 10.1056/NEJMoa067731. Epub 2007 Feb 12. PMID 17296821
- [Result] Lansky AJ, Popma JJ, Cutlip D, Ho KK, Abizaid AS, Saucedo J, Zhang Y, Senerchia C, Kuntz RE, Leon MB, Baim DS. Comparative analysis of early and late angiographic outcomes using two quantitative algorithms in the Balloon versus Optimal Atherectomy Trial (BOAT). Am J Cardiol. 1999 Jun 15;83(12):1611-6. doi: 10.1016/s0002-9149(99)00166-6. PMID 10392863
- [Derived] Gutierrez-Chico JL, Wykrzykowska J, Nuesch E, van Geuns RJ, Koch KT, Koolen JJ, di Mario C, Windecker S, van Es GA, Gobbens P, Juni P, Regar E, Serruys PW. Vascular tissue reaction to acute malapposition in human coronary arteries: sequential assessment with optical coherence tomography. Circ Cardiovasc Interv. 2012 Feb 1;5(1):20-9, S1-8. doi: 10.1161/CIRCINTERVENTIONS.111.965301. Epub 2012 Feb 7. PMID 22319063
- [Derived] Gutierrez-Chico JL, van Geuns RJ, Koch KT, Koolen JJ, Duckers H, Regar E, Serruys PW. Paclitaxel-coated balloon in combination with bare metal stent for treatment of de novo coronary lesions: an optical coherence tomography first-in-human randomised trial, balloon first vs. stent first. EuroIntervention. 2011 Oct 30;7(6):711-22. doi: 10.4244/EIJV7I6A114. PMID 21986329